CLINICAL TRIAL: NCT02930707
Title: Efficacy and Safety of Magnesium Sulfate Added to Local Anesthetic in TAP Block for Postoperative Analgesia Following Total Abdominal Hysterectomy.
Brief Title: TAP Block With Magnesium Sulfate Added to Local Anesthetic in Abdominal Hysterectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, lecturer of anesthesia,ICU, and pain management, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 177
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Pain
Keywords: magnesium sulfate; postoperative pain; TAP block; total abdominal hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Magnesium Sulfate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Magnesium group (Active Comparator): patients received ultrasound guided TAP block with 20 mL of 0.25% bupivacaine plus 2 mL magnesium sulphate 10% (200 mg), on each side of the abdominal wall.
  Interventions: Drug: Magnesium Sulfate
- control group (Placebo Comparator): patients received ultrasound guided TAP block with 20 mL of 0.25% bupivacaine on each side of the abdominal wall.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Magnesium Sulfate — ultrasound guided TAP block with 20 mL of 0.25% bupivacaine plus 2 mL magnesium sulfate 10% (200 mg), on each side of the abdominal wall.
  Arms: Magnesium group
Drug: Bupivacaine — ultrasound guided TAP block with 20 mL of 0.25% bupivacaine on each side of the abdominal wall.
  Arms: control group

SUMMARY:
Major abdominal surgeries are associated with severe abdominal pain, which can affect respiratory and cardiac functions, if insufficiently managed. This increases the incidence of post-operative morbidity.

The objective of this study was to detect the efficacy and safety of magnesium sulphate as an adjuvant to the analgesia offered by local anesthetic in ultrasound guided TAP block in patients undergoing total abdominal hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* weight: 50- 85 kg.
* ASA score: I-III
* scheduled for total abdominal hysterectomy

Exclusion Criteria:

* history of relevant drug allergy.
* coagulation disorders.
* opioid dependence.
* sepsis.
* psychiatric illnesses that would interfere with perception and assessment of pain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
total postoperative morphine consumption | postoperative 24 hours
  total amount of rescue morphine consumption in the first 24 hours postoperatively

SECONDARY OUTCOMES:
postoperative pain | postoperative 24 hours
  postoperative pain measured by VAS score recorded in the first 24 hours postoperatively
first request of rescue analgesia | postoperative 24 hours
  time to the first requirement of rescue analgesia during the first 24 hours postoperatively
side effects | postoperative 24 hours
  occurrence of side effects during the first 24 hours postoperatively

REFERENCES:
- [Derived] Abd-Elsalam KA, Fares KM, Mohamed MA, Mohamed MF, El-Rahman AMA, Tohamy MM. Efficacy of Magnesium Sulfate Added to Local Anesthetic in a Transversus Abdominis Plane Block for Analgesia Following Total Abdominal Hysterectomy: A Randomized Trial. Pain Physician. 2017 Nov;20(7):641-647. PMID 29149143